CLINICAL TRIAL: NCT02001285
Title: Comparison of the Effect-site Concentration of Remifentanil for Blunting Hemodynamic Responses to Ordinary Tracheal and Double-lumen Endobronchial Intubation During Propofol-remifentanil Total Intravenous Anesthesia
Brief Title: Effect-site Concentration of Remifentanil for Blunting Hemodynamic Responses to Double-lumen Endobronchial Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jeju National University School of Medicine (Other)
Responsible Party: Principal Investigator, Hyun Jung Kim, Assistant professor, Jeju National University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HJKim2
Record Dates: First submitted 2013-10-28; First posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Intubation, Intratracheal
Keywords: remifentanil
MeSH Terms: interventions — Remifentanil

ARMS (2):
- Double lumen tube (Experimental): This arm contains patients who are needed endobronchial intubation with double lumen tube for general anesthesia. After propofol infusion of effect site concentration 4 μg/ml, remifentanil infusion will be started with effect site concentration of 3.5 ng/ml. According to change arterial blood pressure and heart rate from baseline value, next remifentanil concentration will be regulated using up-and-down method. Step size of dose is 0.5 ng/ml.
  Interventions: Drug: Remifentanil
- single lumen tube (Active Comparator): This arm contains patients who are needed endotracheal intubation with single lumen tube for general anesthesia. After propofol infusion of effect site concentration 4 μg/ml, remifentanil infusion will be started with effect site concentration of 3.5 ng/ml. According to change arterial blood pressure and heart rate from baseline value, next remifentanil concentration will be regulated using up-and-down method. Step size of dose is 0.5 ng/ml.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — During intubation, remifentanil will be infused to prevent change arterial blood pressure and heart rate.
  Other Names: Ultiva (TM)

SUMMARY:
The purpose of this study is the comparison of the effect-site concentration of remifentanil for blunting hemodynamic responses to ordinary tracheal and double-lumen endobronchial intubation during propofol-remifentanil total intravenous anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient who is needed intubation for general anesthesia

Exclusion Criteria:

* patient who is anticipating difficult airway
* patient who takes any drug to influence this study
* cardiovascular disease, renal disease, liver disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
arterial blood pressure | Change from baseline in arterial blood pressure at intubation period
  Arterial blood pressure will be recorded before anesthesia, after propofol infusion, after remifentanil infusion and after intubation during 3 min with 1 min interval.

SECONDARY OUTCOMES:
heart rate | Change from baseline in heart rate at intubation period
  Heart rate will be recorded before anesthesia, after propofol infusion, after remifentanil infusion and after intubation during 3 min with 1 min interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Jeju National University Hospital, Jeju City, Jeju Special Self-Governing Province, South Korea